CLINICAL TRIAL: NCT05717946
Title: The Influence of Probiotic Supplementation on the Severity of Anxiety and Depressive Symptoms, as Well as the Function and Composition of Gut Microbiota, Metabolic, Inflammation, and Oxidative Stress Markers in Patients With Depression
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Dominik Strzelecki, Professor, MD, PhD, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MULodzAff_1
Record Dates: First submitted 2023-01-06; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Depression; Anxiety
Keywords: probiotics; depression; anxiety; microbiome; metabolism
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, placebo-controlled, and double-blind trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind trial, independent researcher is responsible for randomization and blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I "PRO-D" (Experimental): 50 patients with diagnosed depressive disorders, meeting the criteria of International Classification of Diseases (ICD-11) for 6A70-73, 6A7Y, 6A7Z, taking a probiotic composed of two bacteria strains: Lactobacillus helveticus Rosell and Bifidobacterium longum Rosell.
  Interventions: Dietary Supplement: Probiotic composed of two bacteria strains: Lactobacillus helveticus Rosell and Bifidobacterium longum Rosell.
- Group II "PLC-D" (Placebo Comparator): 50 patients with diagnosed depressive disorders, meeting the criteria of International Classification of Diseases (ICD-11) for 6A70-73, 6A7Y, 6A7Z, taking a placebo.
  Interventions: Other: control group

INTERVENTIONS:
Dietary Supplement: Probiotic composed of two bacteria strains: Lactobacillus helveticus Rosell and Bifidobacterium longum Rosell. — We plan to investigate the impact of the Lactobacillus helveticus Rosell and Bifidobacterium longum Rosell on clinical and biochemical parameters in the experimental group.
  Arms: Group I "PRO-D"
Other: control group — We plan to investigate the impact of a placebo on clinical and biochemical parameters in the control group.
  Arms: Group II "PLC-D"

SUMMARY:
The aim of this study is to gather empirical evidence which will enable to evaluate the impact of probiotic supplementation on the severity of anxiety and depressive symptoms, function, and composition of gut microbiota, metabolic parameters, inflammation, and oxidative stress markers in patients with diagnosed depressive disorders.

The designed study will be prospective, randomized, placebo-controlled, and double-blind. The intervention period will last 8 weeks for each patient. The study will be conducted on 100 patients in total, who will be randomly divided into two groups, consisting of 50 patients each.

Patients included in Group I (PRO-D) will receive one capsule daily containing a probiotic mixture at a daily dose of 3×109 colony-forming units (CFU). The probiotic will be composed of two bacteria strains: Lactobacillus helveticus Rosell®-52, Bifidobacterium longum Rosell®-175, and excipients: potato starch, magnesium stearate, and the capsule shell, made of hydroxypropylmethylcellulose.

Patients included in Group II (PLC-D) will receive daily the same capsule, containing only excipients: potato starch, maltodextrin, and the capsule shell. The color, smell, and taste of the placebo will not be different from those included in the probiotic capsule.

Patients will be considered compliant if they consume >= 80% of the supplements.

The primary outcome measures will be the severity of depressive anxiety and stress symptoms assessed with Montgomery-Åsberg Depression Rating Scale (MADRS) and the Depression, Anxiety, Stress Scale (DASS) with subscales scores, the quality of life level assessed with the WHOQOL-BREF instrument. The secondary outcomes measures will include: blood pressure (BP), body mass index (BMI) and waist circumference (WC) measures, fasting glucose (fGlc), HDL cholesterol (HDL-C), triglycerides (TG), white blood cells count (WBC), neutrofiles, serum levels of C-reactive protein (CRP), the level of faecal SCFAs, faecal microbiota α-diversity and the level of oxidative stress parameters (total antioxidant capacity (TAC) and malondialdehyde (MDA)) in the blood serum.

ELIGIBILITY:
Inclusion Criteria:

1. Depressive disorders diagnosed according to ICD-11,
2. Age between 18 - 70 years,
3. MADRS score >=13,
4. Antidepressant and antianxiety medications not changed 3 weeks prior to the recruitment visit.

Exclusion Criteria:

1. Pregnancy,
2. An infection/vaccination and/or treatment with antibiotics in the previous 4 weeks,
3. Supplementation with pro- or prebiotics in the previous 4 weeks,
4. Having a diagnosis of autoimmune, serious immunocompromised, inflammatory bowel diseases, cancer, IgE-dependent allergy, or severe kidney failure in the previous 4 weeks,
5. body mass index (BMI)> 35,
6. glomerular filtration rate (GFR)< 30 ml/min/1,72 m2,
7. unstable thyroid dysfunction (TSH < 0,27 or > 4,2 μIU/ml) in the previous 4 weeks,
8. Psychiatric comorbidities (except specific personality disorder, additional specific anxiety disorder, and caffeine, and nicotine addiction),
9. Regular treatment (more than 3 days a week) with PPIs, metformin, laxatives, systemic steroids, or NSAIDs in the previous 4 weeks,
10. Significant change in dietary pattern in the previous 4 weeks,
11. Significant change in daily physical activity or extreme sports activity in the previous 4 weeks,
12. Significant change in dietary supplementation in the previous 4 weeks,
13. Significant change in smoking pattern in the previous 4 weeks,
14. High risk of suicide,
15. Is participating in, or has recently participated in, another research study involving an intervention that may alter outcomes of interest to this study,
16. Any other condition or situation which, in the view of investigators, would affect the compliance or safety of the individual taking part.

Reasons for the participant to be discontinued from the study:

1. Withdrawal of informed consent,
2. An infection/vaccination and/or treatment with antibiotics during the trial,
3. Consuming any other than studied probiotics during the trial,
4. Lack of compliance with the probiotic supplementation,
5. Any change in the drug regimen during the study,
6. Exclusion criteria found after enrolment,
7. Any serious adverse event during the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) | 8 weeks
  10-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disturbances. The overall score ranges from 0 to 60 (most severe depression).
Depression, Anxiety, Stress Scale (DASS21) | 8 weeks
  21-item self-administered questionnaire, designed to measure the magnitude of three negative emotional states: depression, anxiety, and stress. These scores ranged from 0 ("did not apply to me at all") to 3 ("apply to me very much or most of the time").
The World Health Organization quality of life-BREF questionnaire (WHOQOL-BREF) | 8 weeks
  6-item questionnaire evaluating four domains: physical health, psychological health, social relationships, and environment validated for several countries.

SECONDARY OUTCOMES:
Blood pressure (BP) | 8 weeks
  Routine measurements in a seated position after 5 minutes of rest.
Body mass index (BMI) | 8 weeks
  Defined as the body mass (kg) divided by the square of the body height (m). Major adult BMI classifications are underweight (under 18.5 kg/m2), normal weight (18.5 to 24.9), overweight (25 to 29.9), and obese (30 or more).
Waist circumference (WC) | 8 weeks
  Wrapping the tape measure around the widest part of stomach, across the navel.
White blood cells count (WBC) | 8 weeks
  The collection will be performed under conditions of fasting, upon overnight resting, in the morning, between 8:00 and 10:00 a.m
Neutrofiles count | 8 weeks
  The collection will be performed under conditions of fasting, upon overnight resting, in the morning, between 8:00 and 10:00 a.m
Serum levels of C-reactive protein (CRP) | 8 weeks
  The collection will be performed under conditions of fasting, upon overnight resting, in the morning, between 8:00 and 10:00 a.m
The level of faecal short-chain fatty acids (SCFAs) | 8 weeks
  Each patient included in the study will be asked to collect a sample of feces twice in a specially designed double sealed bag, which will allow keeping anaerobic conditions.
Faecal microbiota α-diversity | 8 weeks
  Each patient included in the study will be asked to collect a sample of feces twice in a specially designed double sealed bag, which will allow keeping anaerobic conditions.
Total antioxidant capacity (TAC) in the blood serum | 8 weeks
  The collection will be performed under conditions of fasting, upon overnight resting, in the morning, between 8:00 and 10:00 a.m
Malondialdehyde (MDA) level in the blood serum | 8 weeks
  The collection will be performed under conditions of fasting, upon overnight resting, in the morning, between 8:00 and 10:00 a.m
Fasting glucose (fGlc) | 8 weeks
  The collection will be performed under conditions of fasting, upon overnight resting, in the morning, between 8:00 and 10:00 a.m
HDL cholesterol (HDL-C) | 8 weeks
  The collection will be performed under conditions of fasting, upon overnight resting, in the morning, between 8:00 and 10:00 a.m
Triglycerides (TG) | 8 weeks
  The collection will be performed under conditions of fasting, upon overnight resting, in the morning, between 8:00 and 10:00 a.m

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Strzelecki, MD, PhD, Principal Investigator — Medical University of Lodz
Locations (1):
- Central Teaching Hospital, Medical University of Lodz, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Yes
We will publish the study protocol and results with IPD
Supporting Information: Study Protocol
Time Frame: After the publication of both, the study protocol and results.
Access Criteria: open access